CLINICAL TRIAL: NCT01356134
Title: Vascular Fundus Changes in Patients With High Probability of CCSVI (Chronic Cerebrospinal Venous Insufficiency)
Brief Title: Vascular Fundus Changes in Patients With High Probability of Chronic Cerebrospinal Venous Insufficiency (CCSVI)
Status: Completed | Type: Observational
Sponsor: Genetic Disease Investigators (Other)
Collaborators: Optos, PLC (Industry)
Responsible Party: Principal Investigator, Diana Driscoll, O.D., Principal Investigator, Genetic Disease Investigators
Other Study IDs: 61/3527
Record Dates: First submitted 2011-05-12; First posted 2011-05-19 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Ehlers-Danlos Syndrome; Multiple Sclerosis
Keywords: multiple sclerosis; ehlers danlos syndrome; CCSVI; chronic cerebrospinal venous insufficiency; fundus; retina
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Multiple sclerosis and or Ehlers-Danlos: Patients with suspected or confirmed cases of Ehlers Danlos Syndrome and or Multiple Sclerosis
- Age matched normals: Age matched normals

SUMMARY:
The investigators propose that evidence of chronic cerebrospinal venous insufficiency (CCSVI) may be evident in the vasculature of the fundus. The investigators will be examining fundi of multiple sclerosis patients and Ehlers-Danlos patients to see if evidence of CCSVI can be found in these patients having high risk for CCSVI. The investigators will read the fundus photos, compared to age-matched normals in a "blind" fashion.

DETAILED DESCRIPTION:
Chronic Cerebrospinal Venous Insufficiency (CCSVI) has been proposed as the cause of numerous neurodegenerative diseases of the brain. CCSVI is the result of poor drainage of blood (and cerebral spinal fluid to some degree) from weakened or stenosed veins usually located in the cervical area (most notably the internal jugular veins). Although current focus and treatment of CCSVI is on multiple sclerosis, CCSVI has also been implicated as a potential cause of Alzheimer's disease and Parkinson's Disease. Additionally, patients with Ehlers-Danlos Syndrome (EDS) -- a disorder of connective tissue -- are more prone to developing multiple sclerosis than the general population. Many EDS patients are known to have weakened and abnormal blood vessels and 40 - 70% of EDS patients develop autonomic dysfunction in addition to numerous other symptoms found in patients with CCSVI. In the small subset of EDS and multiple sclerosis patients seen at Total Eye Care, the investigators have noticed a vascular irregularity (using the optomap® and examining the results under high magnification) which offers credence to the theory of CCSVI. Such objective data has been elusive, excepting for fMRI, ultrasound (to a limited degree) and venous angioplasty results. Current treatment of CCSVI involves the ballooning and sometimes stenting, of abnormally stenosed veins. The treatment of CCSVI offers hope to many patients suffering from multiple sclerosis. Although CCSVI research is in its infancy, many doctors believe that CCSVI is a significant portion of the solution to patients with neurodegenerative diseases of the brain. Because CCSVI is a vascular disorder, the investigators hypothesize that the investigators are able to screen candidates for CCSVI via the optomap®.

ELIGIBILITY:
Inclusion Criteria:

* age matched normals
* patients with diagnosed or suspected Ehlers-Danlos Syndrome and/or diagnosed or suspected Multiple Sclerosis ("CIS")

Exclusion Criteria:

* diabetics and patients unable to sit in position for testing are excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Aged-matched normals are patients at Total Eye Care. Multiple sclerosis and/or Ehlers-Danlos patients will be accepted from any area, and will not be excluded based on location of residence. They need not be patients of Total Eye Care.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Fundus: venous engorgement/beading | Baseline
  Abnormal vessel appearance in fundi may include venous engorgement and beading, abnormal A/V ratio, blurred disc margins, papilledema, dot hemorrhages or exudates.

CONTACTS AND LOCATIONS:
Overall Officials: Diana L Driscoll, O.D., Study Director — Genetic Disease Investigators; Richard A Driscoll, O.D., Principal Investigator — Genetic Disease Investigators; Clair A Francomano, M.D., Study Chair — Harvey Institute for Human Genetics
Locations (1):
- Total Eye Care, Colleyville, Texas, United States

REFERENCES:
- [Background] Vilisaar J, Harikrishnan S, Suri M, Constantinescu CS. Ehlers-Danlos syndrome and multiple sclerosis: a possible association. Mult Scler. 2008 May;14(4):567-70. doi: 10.1177/1352458507083187. Epub 2008 Jan 21. PMID 18208891
- [Background] Singh AV, Zamboni P. Anomalous venous blood flow and iron deposition in multiple sclerosis. J Cereb Blood Flow Metab. 2009 Dec;29(12):1867-78. doi: 10.1038/jcbfm.2009.180. Epub 2009 Sep 2. PMID 19724286
- [Background] Zamboni P, Galeotti R, Menegatti E, Malagoni AM, Tacconi G, Dall'Ara S, Bartolomei I, Salvi F. Chronic cerebrospinal venous insufficiency in patients with multiple sclerosis. J Neurol Neurosurg Psychiatry. 2009 Apr;80(4):392-9. doi: 10.1136/jnnp.2008.157164. Epub 2008 Dec 5. PMID 19060024